CLINICAL TRIAL: NCT05608785
Title: Single-center, Multi-cohort Exploratory Phase Ib/II Clinical Study of First-line Treatment of Unresectable Locally Advanced/Advanced Adenocarcinoma of the Stomach or Gastroesophageal Junction Based on Different Genotypes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-MATCH
Record Dates: First submitted 2022-09-15; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer; Gastroesophageal-junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HER2 protein positive 3+ or FISH amplification or HER protein 2+ but FISH amplification (Experimental): Initial treatment (4-6 cycles): IBI315 injection, oxaliplatin, capecitabine
  * IBI315: 1200 mg per cycle d1 dosing, intravenous drip, 3 weeks as one treatment cycle.
  * Oxaliplatin: 130 mg/m2, d1 per cycle, intravenous drip, 3 weeks as a treatment cycle.
  * Capecitabine: 1000 mg/m2 orally twice daily (1 dose in the morning and 1 dose in the evening), d1-d14 per cycle, 2 weeks off 1 week, 3 weeks cycle.
  Patients with CR/PR/SD enter maintenance therapy: IBI315 monotherapy maintenance
  - IBI315: 1200 mg IV drip per cycle d1 for 3 weeks.
  Interventions: Drug: IBI315; Drug: Oxaliplatin; Drug: Capecitabine
- Positive for Claudin 18.2 protein (Experimental): Initial treatment (4-6 cycles): PD-L1 monoclonal antibody, TST001 injection, oxaliplatin, capecitabine
  * TST001: 3mg, 4.5mg and 6mg dose levels for hill climbing trial, dose per cycle d1, IV drip, 3 weeks for one treatment cycle. 3-6 patients were enrolled in each dose level (3 patients were enrolled if no DLT was present, if present extended to 6 patients)
  * TQB2450 injection: 1200 mg per cycle d1 dosing, IV drip, 3 weeks as a treatment cycle.
  * Oxaliplatin: 130 mg/m2 per cycle d1 dosing, intravenous drip, 3 weeks as a treatment cycle.
  * Capecitabine: 1000 mg/m2 orally twice daily (1 dose in the morning and 1 dose in the evening), d1-d14 per cycle, 2 weeks off 1 week, 3 weeks cycle.
  Patients with CR/PR/SD enter maintenance therapy: TQB2450 injection + TST001
  * TST001: maintenance at the dose level used (3mg/4.5mg/6mg), dosed d1 per cycle, IV drip, 3 weeks as a treatment cycle.
  * TQB2450 injection: 1200mg, dosed d1 per cycle, intravenous drip, 3 weeks as a treatment cycle.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: TST001; Drug: TQB2450
- Her2 protein, Claudin18.2 protein were negative (Experimental): Initial treatment (4-6 cycles): TQB2450 injection, Anrotinib, Oxaliplatin, Capecitabine
  * TQB2450 injection: 1200mg per cycle d1 dosing, intravenous drip, 3 weeks as a treatment cycle.
  * Anrotinib: 1 capsule (10 mg) once daily, dosed every cycle d1-d14, stopping for 2 consecutive weeks, 3 weeks as a treatment cycle
  * Oxaliplatin: 130 mg/m2, d1 per cycle, intravenous drip, 3-week treatment cycle.
  * Capecitabine: 1000 mg/m2 orally twice daily (1 dose in the morning and 1 dose in the evening), d1-d14 per cycle, 2 weeks off 1 week, 3 weeks as a treatment cycle.
  Patients with CR/PR/SD enter maintenance therapy: PD-L1 inhibitor, anlotinib
  * PD-L1 monoclonal antibody (TQB2450): 1200 mg d1 per cycle, intravenous drip, 3 weeks as a treatment cycle.
  * Anlotinib: 1 capsule (10mg) once daily, d1-d14 per cycle, stopping for 2 weeks, 3 weeks as a treatment cycle.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: TQB2450; Drug: Anrotinib

INTERVENTIONS:
Drug: IBI315 — IBI315 is a recombinant fully humanized anti-programmed death receptor 1 (PD-1) and humanized anti-human epidermal growth factor receptor 2 (HER2) bispecific antibody injection.
  Arms: HER2 protein positive 3+ or FISH amplification or HER protein 2+ but FISH amplification
Drug: Oxaliplatin — Oxaliplatin is a type of chemotherapy. It is used as a treatment for different types of cancer, including gastric cancer.
Drug: Capecitabine — Capecitabine is a type of chemotherapy. It is used as a treatment for different types of cancer, including gastric cancer.
Drug: TST001 — TST001 is a high-affinity humanized monoclonal antibody targeting Claudin 18.2 with enhanced antibody-dependent cytotoxic (ADCC) and complement-dependent cytotoxic (CDC) activity, showing potent antitumor activity in xenograft assays.
  Arms: Positive for Claudin 18.2 protein
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
  Arms: Her2 protein, Claudin18.2 protein were negative; Positive for Claudin 18.2 protein
Drug: Anrotinib — Anlotinib is a novel multitarget tyrosine kinase inhibitor for tumor angiogenesis and proliferative signaling.
  Arms: Her2 protein, Claudin18.2 protein were negative

SUMMARY:
Abstract Study title: Single-center, Multi-cohort Exploratory Phase Ib/II Clinical Study of First-line Treatment of Unresectable Locally Advanced/Advanced Adenocarcinoma of the Stomach or Gastroesophageal Junction Based on Different Genotypes Protocol No: GC-MATCH Initiator: Henan Cancer Hospital Nature of study Investigator-initiated exploratory study Subjects Advanced first-line gastric cancer or adenocarcinoma of the gastroesophageal junction Objective: To evaluate the efficacy and safety of different first-line treatment options for unresectable locally advanced/advanced gastric or combined gastroesophageal adenocarcinoma with different gene/protein types.

Evaluation criteria: To evaluate the adverse effects of drugs using the NCI CTCAE V5.0 criteria.

RECIST1.1 criteria were used to evaluate drug efficacy Study endpoints: Primary indicators Objective Response Rate (ORR) Secondary indicators 1. drug safety. 2. disease control rate DCR (CR+PR+SD). 3. duration of remission DoR. 4. disease-free survival (PFS) and overall survival time (OS). 5. R0/R1 surgical resection rate Study design: Single-center umbrella clinical trial Planned number of enrollment: Total 39-45 cases Sample size estimation: This is an exploratory study and sample size was not calculated Statistical methods: Selection of data for statistical analysis Full Analysis Set (FAS): The efficacy analysis was performed on all patients who were enrolled and used the drug at least once, according to the principle of intentional analysis (ITT).

Per-protocol Set: Cases with at least one oncologic efficacy assessment, compliance with the trial protocol, good compliance, no prohibited drugs during the trial, and completion of the case report form.

Safety Analysis Set: All patients who had used the trial drug at least once and had a safety record after the drug was administered were enrolled in the Safety Analysis Set.

Statistical analysis plan Validity analysis: for the efficacy index PFS, the Kaplan-Meier method will be used to estimate its median time and column Statistical methods: Out of two-sided 95% confidence intervals. Disease control rate (DCR = CR+PR+SD) and objective remission rate (ORR = CR+PR) were calculated using Fisher exact probability and bilateral 95% confidence intervals were presented.

Safety analysis: descriptive statistical analysis was used to tabulate the AEs that occurred in this trial. laboratory test results were described as normal before the trial but abnormal after treatment and in relation to the trial drug when abnormal changes occurred.

Treatment protocol:

All subjects in this study were first tested for genes/proteins (HER2 protein, HER2FISH, PD-L1 protein 22C3, Claudin18.2, MMR) and received treatment in different groups according to gene/protein expression.

Group 1 HER protein positive 3+ or FISH amplification or HER protein 2+ but FISH amplification Initial treatment (4-6 cycles): IBI315 injection, oxaliplatin, capecitabine Group 2 Claudin18.2 protein-positive Initial treatment (4-6 cycles): PD-L1 monoclonal antibody, TST001 injection, oxaliplatin, capecitabine Group 3 Her protein and Claudin18.2 protein were negative Initial treatment (4-6 cycles): TQB2450 injection, Anrotinib, Oxaliplatin, Capecitabine Patients can undergo radical gastric cancer surgery or radical gastric cancer surgery + local treatment during the maintenance treatment phase if their condition is stable and after in-hospital MDT consultation. The duration of maintenance treatment was 2 years from the time of enrollment.

Principal Investigator: Luo Suxia, Li Ning Group leader unit: Henan Cancer Hospital

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form for this study.
* Male or female patients aged 18-75 years.
* unresectable advanced or metastatic gastric cancer or adenocarcinoma of the gastroesophageal junction (including indolent cell carcinoma, mucinous adenocarcinoma, hepatoid adenocarcinoma) confirmed by pathological (histological or cytological) examination.
* >6 months from the end of prior (neo)adjuvant chemotherapy/adjuvant radiotherapy to the time of disease recurrence
* at least one measurable lesion or evaluable lesion according to RECIST version 1.1; measurable lesions should not have received local treatment such as radiotherapy (lesions located within the area of previous radiotherapy may also be optional targets if progression is confirmed and they meet RECIST 1.1 criteria)
* ECOG score: 0 to 1.
* Life expectancy ≥ 3 months.
* Adequate organ function, with the following laboratory test values required at screening.
* Routine blood test criteria to be met. Hemoglobin level (HB) ≥ 90 g/L (no blood transfusion within 14 days). Absolute neutrophil count (ANC) ≥ 1.5 x 109/L. Platelet count (PLT) ≥100×109/L (no interleukin 11 or TPO within 14 days). White blood cell count (WBC) ≥4.0×109/L (no granulocyte stimulating factor within 14 days).
* Biochemical tests are required to meet the following criteria. Serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN). ALT and AST ≤ 2.5 ULN. Cr ≤ 1.5 ULN or creatinine clearance (CCr) ≥ 60 ml/min, (Cockcroft-Gault formula).

Serum albumin ≥ 25 g/L (2.5 g/dL). For subjects with liver metastases, AST and ALT must be ≤ 5 x ULN, leukocytes ≥ 4 x 109/L, untransfused platelets ≥ 100 x 109/L, absolute neutrophil value (ANC) without granulocyte-stimulating factor treatment ≥ 1.5 x 109/L, hemoglobin ≥ 90 g/L

* Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ low limit of normal (50%).
* Adequate coagulation, defined as an international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN.
* Women of childbearing potential are required to use highly effective contraception for the duration of the study, and for the period after the last dose and for at least 180 days after chemotherapy. It is recommended that contraception be initiated at least 3 months prior to study drug administration; non-sterile men are required to use highly effective contraception for the duration of the study and for at least 180 days after both the last dose and chemotherapy. It is recommended that contraception be initiated at least 3 months prior to study drug administration.
* If local treatment of metastases, such as radiotherapy or ablation, is performed, they may also be enrolled after 14 days of washout as long as an assessable lesion is still present and the local treatment is not followed by anti-tumor therapy such as targeted, chemotherapy or immunotherapy.

Exclusion Criteria:

* Hypersensitivity to any of the test drugs and their excipients, or a history of severe allergy, or a contraindication to the test drug.
* A history or active stage of autoimmune disease.
* symptomatic/asymptomatic brain metastases
* CT suggestive of definite ulcerative lesions or positive fecal occult blood (risk of bleeding and suitability for enrollment as determined by the investigator)
* History of abnormal bleeding (except epistaxis) complained of 14 days prior to enrollment
* previous allogeneic bone marrow transplantation or organ transplantation
* congenital pulmonary fibrosis, drug-induced pneumonia, mechanized pneumonia, or CT-confirmed active pneumonia
* HIV positive test, active hepatitis B or C, active tuberculosis.
* Uncontrolled cancer pain.
* previous live attenuated vaccine within 4 weeks prior to study entry or expected to be administered during or within 5 months of the end of the trial
* Prior treatment with PD-1/PD-L1 antibodies, CTLA-4 antibodies, or other therapies targeting PD-1/PD-L1 and/or VEGFR inhibitors or have not recovered from adverse events caused by dosing >4 weeks prior (i.e., have not returned to ≤ grade 1 or baseline levels)).
* Systemic application of glucocorticoids or immunosuppressants within 2 weeks prior to trial start (note: inhaled glucocorticoids and salicorticoids are permitted).
* Known presence of symptomatic CNS metastases and/or carcinomatous meningitis. Patients with a history of CNS metastases or spinal cord compression may be enrolled in the study if they are clearly treated and clinically stable after discontinuation of anticonvulsants and steroids for 4 weeks prior to the first dose of the study.
* Have a contraindication to hormone use.
* Have multiple factors that interfere with oral drug administration (e.g., inability to swallow, chronic diarrhea, and intestinal obstruction)
* peripheral neuropathy ≥ NCI CTCAE grade 2.
* Uncontrollable or symptomatic hypercalcemia.
* infections requiring antibiotics within 14 days prior to the start of the trial
* chronic enterocolitis.
* Patients with bone metastases at risk of paraplegia.
* Patients with any severe and/ or uncontrolled disease, including: Patients with suboptimal blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg) on antihypertensive medications; patients with class II or higher myocardial ischemia or myocardial infarction, arrhythmias (including QT interval ≥ 480 ms); class III-IV cardiac insufficiency by NYHA criteria, or cardiac ultrasound suggestive of left ventricular ejection fraction ( LVEF) <50% in patients. Active or uncontrolled severe infections. Liver disease such as cirrhosis, decompensated liver disease, chronic active hepatitis. Poorly controlled diabetes mellitus (fasting blood glucose (FBG) >10 mmol/L). Urine routine suggestive of urine protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g.
* Long-term untreated wounds or fractures 23) Subjects who are unable to receive a trans-peripheral central venous placement (PICC)
* Subjects with abnormal coagulation (INR > 1.5 or APTT > 1.5 × ULN), with bleeding tendency or on thrombolytic or anticoagulant therapy. Known hereditary or acquired bleeding and thrombotic tendencies such as: hemophilia, impaired coagulation skills, thrombocytopenia, hypersplenism, etc. Active bleeding within 14 prior to study entry.
* Major surgical procedure (craniotomy, open-heart or open-heart surgery) within 4 weeks prior to the first dose of study, or anticipated need for major surgery during study treatment, or non-diagnostic surgery within 4 weeks prior to the start of the trial.
* history of gastrointestinal perforation and/or fistula within 3 months prior to enrollment in treatment; or arterial/venous thrombotic events such as cerebrovascular accidents (except stable cerebral infarction as assessed by the investigator), deep vein thrombosis, and pulmonary embolism (except if cured)
* Clinically significant thoracoabdominal fluid, including any thoracoabdominal fluid that is detectable on physical examination, previously treated or currently still requiring treatment Those with only a small amount of thoracic ascites on imaging but asymptomatic, which the investigator assesses does not require treatment may be enrolled.
* Interstitial lung disease requiring steroid hormone therapy.
* uncontrolled metabolic disorders or other non-malignant organ or systemic diseases or secondary reactions to cancer that can lead to higher medical risk and/or uncertainty in survival evaluation
* Patients with significant malnutrition.
* Patients with a history of psychotropic substance abuse and inability to abstain or with psychiatric disorders
* those with a history of immunodeficiency, including testing positive for HIV or having other acquired, congenital immunodeficiency disorders, or a history of organ transplantation
* History of other primary malignancies, except for 1) malignancies in complete remission for at least 2 years prior to enrollment and requiring no other treatment during the study period; 2) non-melanoma skin cancers or malignant freckled nevi that have been adequately treated and have no evidence of disease recurrence; and 3) carcinomas in situ that have been adequately treated and have no evidence of disease recurrence.
* Female patients who are pregnant or breastfeeding.
* those who, in the judgment of the investigator, have a serious concomitant disease that jeopardizes patient safety or interferes with the patient's ability to complete the study
* Participating in another trial within 30 days prior to the start of the trial, or planning to participate in another trial while the trial is ongoing.
* Inclusion in the row with the most stringent conditions, if there is duplication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | up to 100 months
  An adverse event contains multiple severity grades, typically the start date is the date of mild (grade 1) occurrence, the end date is the date of improvement, and the level is filled in at the highest level.

SECONDARY OUTCOMES:
Objective response rate，ORR | up to 100 months
  The remission period is usually defined as the period from the onset of efficacy until the confirmation of tumor progression. The objective remission rate is generally defined as the sum of complete remission plus partial remission (CR+PR).
Duration of Response, DoR | up to 100 months
  Time from when the patient first achieved complete remission or partial remission to disease progression.
progression-free survival，PFS | up to 100 months
  Time from randomization grouping of patients to disease progression or death from any cause.
overall survival，OS | up to 100 months
  From date of randomization until the date of death from any cause, assessed up to 100 months
disease control rate，DCR | up to 100 months
  Proportion of patients who achieve complete remission, partial remission, or disease control with optimal efficacy
R0/R1 resection rate | up to 100 months
  R0/R1 resection rate